CLINICAL TRIAL: NCT00529477
Title: The Effects of Methacholine Challenge Administered Using Three Different Nebulizers on Small Airways Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Gail Gauvreau, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NEB3-AIR
Record Dates: First submitted 2007-09-07; First posted 2007-09-14 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): The Wright Nebulizer will be used to perform the methacholine challenge in arm 1.
  Interventions: Other: 1. Wright Nebulizer
- 2 (Active Comparator): The Pari LC nebulizer will be used to perform the methacholine challenge in arm 2.
  Interventions: Other: Pari LC Nebulizer
- 3 (Active Comparator): The Pari Sinustar nebulizer will be used to perform the methacholine challenge in arm 3.
  Interventions: Other: The Pari Sinustar Nebulizer

INTERVENTIONS:
Other: 1. Wright Nebulizer — The Wright nebulizer will be used to perform the methacholine challenge.
  Arms: 1
Other: Pari LC Nebulizer — The Pari LC nebulizer will be used to perform the methacholine challenge.
  Arms: 2
Other: The Pari Sinustar Nebulizer — The Pari Sinustar nebulizer will be used to perform the methacholine challenge.
  Arms: 3

SUMMARY:
The objective of this study is to examine the functional effects of methacholine challenge on small airways using three different nebulizers to generate particles with HMAD suitable for distribution in small, intermediate and large airways.Pulmonary function will be assessed using plethysmography and impulse oscillation techniques. Eight asthmatic subjects (>18 years, both sexes) who are stable clinically and require only intermittent ß2-agonist treatment will be recruited to undergo methacholine challenges for an in vivo, dose-finding observational study. Three separate methacholine challenges will be carried out using each of the three different nebulizers. After each challenge, pulmonary function tests will be performed on subjects to assess functional changes in large and small airways. Results of the tests will be compared between the three nebulizers. These experiments will demonstrate whether or not functional changes occur in small airways in response to methacholine, as measured by pulmonary function tests after selectively targeting small airways using the nebulizer which generates small particles. The results from these experiments will give us a better understanding of the role of small airways in methacholine-induced bronchoconstriction in asthmatics, and will compare sensitivity of plethysmography compared to forced oscillation for detecting changes in small airways.

DETAILED DESCRIPTION:
This study will measure changes in small airways by plethysmography and impulse oscillation following delivery of methacholine using nebulizers designed to deliver to the small (Wright), intermediate (PARI LC® Plus) and large (PARI SinuStar™ ) airways.

Assessment of small airways involvement by plethysmography will include Residual Volume (RV), Forced Vital Capacity (FVC) and Peak Inspiratory and Expiratory Flow rates (PIF and PEF, respectively). Impulse oscillation will include measures of large and small airways resistance.

Baseline Spirometry

Baseline FEV1 and VC will be registered using a water spirometer.

Methacholine Challenge (Screening)

Methacholine inhalation will be performed as described by Cockcroft (1996). Subjects are instructed to wear noseclips and to breathe normally from the mouthpiece during the 2-minute inhalation period. Subjects inhale normal saline, then doubling concentrations of methacholine from a Wright nebulizer for 2 minutes each. FEV1 is measured at 30, 90, 180 and 300 seconds after each inhalation. Spirometry is measured with a Collins water sealed spirometer and kymograph. The test is terminated when a fall in FEV1 of 20% of the baseline value occurs, and the methacholine PC20 is calculated.

Methacholine Challenge

During the second visit, subjects will be randomized to inhale from a nebulizer that generates particles with HMAD suitable for distribution either in small, intermediate or large airways. Subjects will inhale doubling concentrations of methacholine for 2 minutes each. Immediately after each inhalation, pulmonary function tests will be performed on the subjects via plethysmography. Measurements will be made at intervals of 30 seconds, 60 seconds, 3 minutes and 5 minutes (or until a fall in FEV1 of 20% or more of baseline is reached). The methacholine test is terminated when a fall in FEV1 of 20% or more of the baseline value is reached. After a recovery time of 1 hour, the same doses will be re-administered and pulmonary function tests will again be performed, this time via impulse oscillation. The same procedure will be repeated for the third and fourth visits with the remaining nebulizers (selected randomly). The nebulizers that will be used to target certain airways are the Wright nebulizer (small), the PARI LC® Plus nebulizer (medium) and the PARI SinuStar™ nebulizer (large).

Plethysmography

Pulmonary function tests will be performed on subjects after methacholine challenges via plethysmography. Various tests will be performed that will allow for different lung function measures. To characterize which measurements are indicative of large or small airways function, measurements from the three nebulizer groups will be compared. Potential measures of small airway function include Functional Residual Capacity (FRC), Residual Volume (RV), Forced Vital Capacity (FVC) and Peak Inspiratory and Expiratory Flow Rates (PIF and PEF, respectively) (Knudson et al., 1980). Nitrogen washout will also be performed with the body box to measure airway distensibility, or the relationship between airway caliber and lung volume (Brown et al., 2004).

Impulse Oscillation

Pulmonary function tests will be performed on subjects after methacholine challenges via impulse oscillation. This device uses a loudspeaker to generate pressure and flow and by generating these at various frequencies, specifically differentiates between large and small airways obstruction (Otis et al., 1956). Results will be compared between the three nebulizer groups after specifically targeting certain airways.

ELIGIBILITY:
Inclusion Criteria:

* Mild asthmatics, presently well controlled on ß2-agonists.
* Non-smokers.
* Baseline FEV1 more than 70% of predicted normal.

Exclusion Criteria:

* Airway infection during the last 4 weeks.
* Exacerbation during the last 4 weeks.
* Inhaled or oral steroids during the last 4 weeks.
* Antihistamines during the last 48 hours.
* Asthma medication other than inhaled and/or oral ß2-agonists during the last 4 weeks.
* Pregnant women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To examine the functional effects of methacholine challenge on small airways via plethysmography and impulse oscillation techniques | April 2008
To compare the sensitivity of these measurement techniques to detect changes in small airways. | April 2008

CONTACTS AND LOCATIONS:
Overall Officials: Kieran Killian, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Naji N, Keung E, Beaudin S, Kane J, Killian KJ, Gauvreau GM. The effects of particle size on measurement of airway hyperresponsiveness to methacholine. Ann Allergy Asthma Immunol. 2013 May;110(5):359-63. doi: 10.1016/j.anai.2013.02.014. Epub 2013 Mar 19. PMID 23622007